CLINICAL TRIAL: NCT06670118
Title: EXPLORING the CORRELATION of the LUNG ULTRASOUND with DELIRIUM and OUTCOMES in ACUTE GERIATRICS WORLD (ECO-AGE): a MULTICENTER, PROSPECTIVE, OBSERVATIONAL STUDY from the GRETA GROUP (GRUPPO DI RICERCA in ECOGRAFIA TORACICA NELL' ANZIANO) of the ITALIAN SOCIETY of GERONTOLOGY and GERIATRICS (SIGG)
Brief Title: Exploring the Correlations of Lung Ultrasound with Delirium and Outcomes in Acute GEriatrics World: a Multicenter, Prospective, Observational Study from the GRETA Group of the Italian Society of Gerontology and Geriatrics
Acronym: ECO-AGE
Status: Not yet recruiting | Type: Observational
Sponsor: University of Milano Bicocca (Other)
Responsible Party: Sponsor
Other Study IDs: ID 4369_20.03.2024_M bis
Record Dates: First submitted 2024-10-31; First posted 2024-11-01 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Acute Respiratory Failure; Delirium in Old Age; Pneumonia; Acute Heart Failure (AHF); Chronic Obstructive Pulmonary Disease (COPD); Ultrasound Exams
Keywords: Lung Ultrasound Abnormalities in Older Adults; Lung ultrasound; delirium; respiratory failure; geriatrics
MeSH Terms: conditions — Pneumonia; Pulmonary Disease, Chronic Obstructive; Delirium; Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients with Normal Lung Ultrasound (LUS) Findings: This cohort includes patients aged 65 and older admitted with acute respiratory symptoms who undergo lung ultrasound (LUS) upon hospital admission. LUS findings in this cohort show normal lung conditions with no significant pleural or parenchymal abnormalities (e.g., no comet-tail artifacts, consolidations, or effusions). The primary interest is to assess the absence of LUS abnormalities and their correlation with clinical outcomes, including delirium, oxygen therapy, and mortality.
- Patients with Abnormal Lung Ultrasound (LUS) Findings: This cohort includes patients aged 65 and older admitted with acute respiratory symptoms who undergo lung ultrasound (LUS) upon hospital admission. LUS findings in this cohort show significant abnormalities such as pleural effusions, consolidations, or diffuse comet-tail artifacts (B-lines). The primary interest is to assess the presence of LUS abnormalities and their correlation with clinical outcomes, including delirium, duration of hospitalization, need for oxygen therapy, non-invasive ventilation, and mortality.

SUMMARY:
The purpose of this observational study is to investigate the prognostic relevance of lung ultrasound (LUS) performed on older patients (aged 65 and above) admitted to the hospital with acute respiratory symptoms. The primary objective is to determine if LUS-detected pulmonary abnormalities upon hospital admission are associated with the development of delirium during hospitalization. Secondary objectives include assessing the association between LUS patterns and clinical outcomes such as oxygen supplementation duration, non-invasive ventilation use, mortality, and length of hospital stay. This study involves no interventions and will monitor patients using LUS as part of their regular clinical care in multiple centers.

DETAILED DESCRIPTION:
This is a multicenter, prospective, observational study designed to explore the prognostic value of lung ultrasound (LUS) in older patients admitted with acute respiratory symptoms. The study, titled "Exploring the Correlations of Lung Ultrasound with Delirium and Outcomes in Acute Geriatrics world (ECO-AGE)," aims to evaluate whether the presence of LUS abnormalities, such as pleural or lung parenchymal changes, detected upon admission is associated with the onset of delirium during hospitalization.

The study will recruit participants aged 65 years or older who are admitted to the hospital through the emergency room due to acute respiratory complaints (e.g., dyspnea, cough, reduced oxygen saturation, clinical suspicion of pneumonia, acute heart failure, or chronic obstructive pulmonary disease). Patients will undergo LUS as part of their routine clinical management, and data collected from the LUS exams will be analyzed to assess correlations with clinical outcomes.

The primary endpoint of the study is the incidence of delirium, measured using the 4AT scale, during the hospital stay. Secondary endpoints include associations between LUS patterns and the following outcomes:

Duration of oxygen therapy Requirement for non-invasive mechanical ventilation Length of hospital stay In-hospital mortality Readmission rates and mortality at 3 months post-discharge The study hypothesizes that certain LUS abnormalities, such as diffuse or focal comet-tail artifacts (B-lines), pleural effusion, or parenchymal consolidations, will be predictive of adverse outcomes like delirium or prolonged respiratory support.

Data will be collected via electronic Case Report Forms (eCRFs) and analyzed using multivariate regression models, adjusting for potential confounders such as age, sex, frailty, and comorbidities. The estimated recruitment period is 12 months, and patient outcomes will be monitored throughout hospitalization and for 3 months following discharge. The findings of this study are expected to inform better risk stratification and clinical management of older patients with acute respiratory illnesses.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 65 years or older, admitted directly from the Emergency Room or Emergency Medical Services with acute respiratory symptoms or signs.

Presence of acute respiratory symptoms, including:

* Dyspnea or cough.
* Oxygen saturation less than 94% or respiratory rate ≥ 22 breaths per minute, or PaO2/FiO2 < 300.
* Clinical suspicion of acute respiratory illness (e.g., pneumonia, acute congestive heart failure, pulmonary edema, COPD, pleural effusion, pneumothorax).
* Lung ultrasound (LUS) performed within 48 hours of admission for clinical reasons.
* Signed informed consent for participation in the study.

Exclusion Criteria:

* Presence of delirium upon admission.
* Refusal to sign the informed consent form or consent to data collection.
* Terminal illness with an estimated survival prognosis of no more than 3 months.
* Previous open thoracic or cardiothoracic surgery compromising the quality of LUS images.
* Lack of cooperation during the LUS examination.
* Any condition determined by the investigators that could introduce bias into the study or compromise the quality of the LUS examination.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The study population will consist of patients aged 65 years and older admitted to participating hospitals through the emergency room or emergency medical services with acute respiratory symptoms (e.g., dyspnea, cough, low oxygen saturation). These patients will undergo lung ultrasound (LUS) as part of their routine clinical management. The study will focus on older adults presenting with conditions such as pneumonia, acute congestive heart failure, chronic obstructive pulmonary disease (COPD), pleural effusion, or pneumothorax. The population will include both male and female patients from multiple centers across Italy, with a particular focus on those at higher risk of delirium and poor clinical outcomes due to underlying frailty or multimorbidity.
Sampling Method: Non-Probability Sample
Enrollment: 480 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Correlation Between LUS-Detected Pulmonary Abnormalities and Delirium Occurrence | During the hospital stay (assessed daily), up to 30 days
  The primary outcome measure is the correlation between lung ultrasound (LUS)-detected pulmonary abnormalities and the occurrence of delirium, assessed daily using the 4AT scale during hospitalization

SECONDARY OUTCOMES:
Correlation Between LUS Characteristics and Duration of Delirium | During the hospital stay (up to 30 days)
  The duration of delirium, measured in days, will be correlated with LUS characteristics. Delirium duration will be evaluated using daily assessments with the 4AT scale.
Correlation Between LUS Characteristics and Duration of Oxygen Administration | During the hospital stay (up to 30 days)
  The correlation between LUS findings and the duration of oxygen therapy, measured in days. Oxygen therapy duration will be tracked throughout hospitalization.
Correlation Between LUS Characteristics and PaO2/FiO2 Ratio | During the hospital stay (up to 30 days)
  The correlation between LUS findings and the ratio of arterial oxygen pressure (PaO2) to fractional inspired oxygen (FiO2), based on blood gas analyses during hospitalization.
Correlation Between LUS Characteristics and Need for Non-Invasive Ventilation (NIV) | During the hospital stay (up to 30 days)
  The correlation between LUS findings and the requirement for non-invasive ventilation (NIV). The need for NIV and the duration of ventilatory support will be recorded.
Correlation Between LUS Characteristics and Duration of Hospitalization | During the hospital stay (up to 30 days)
  The correlation between LUS findings and the duration of hospitalization, measured in days from admission to discharge.
Correlation Between LUS Characteristics and In-Hospital Mortality | During the hospital stay (up to 30 days)
  The correlation between LUS findings and in-hospital mortality. This outcome will include the number of patients who die during hospitalization.
Correlation Between LUS Characteristics and 3-Month Readmission and Mortality Rates | 3 months after discharge
  The correlation between LUS findings and readmission or mortality within 3 months after hospital discharge. Follow-up will be conducted through phone calls to the patients or caregivers.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe GB Bellelli, Medical Doctor, Principal Investigator — University of Milano Bicocca
Locations (1):
- Fondazione IRCCS San Gerardo, Monza, MB, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bellelli G, Brathwaite JS, Mazzola P. Delirium: A Marker of Vulnerability in Older People. Front Aging Neurosci. 2021 Apr 30;13:626127. doi: 10.3389/fnagi.2021.626127. eCollection 2021. PMID 33994990
- [Background] Ormseth CH, LaHue SC, Oldham MA, Josephson SA, Whitaker E, Douglas VC. Predisposing and Precipitating Factors Associated With Delirium: A Systematic Review. JAMA Netw Open. 2023 Jan 3;6(1):e2249950. doi: 10.1001/jamanetworkopen.2022.49950. PMID 36607634
- [Background] Limpawattana P, Phungoen P, Mitsungnern T, Laosuangkoon W, Tansangworn N. Atypical presentations of older adults at the emergency department and associated factors. Arch Gerontol Geriatr. 2016 Jan-Feb;62:97-102. doi: 10.1016/j.archger.2015.08.016. Epub 2015 Aug 21. PMID 26323650
- [Background] Vetrugno L, Guadagnin GM, Barbariol F, Langiano N, Zangrillo A, Bove T. Ultrasound Imaging for Diaphragm Dysfunction: A Narrative Literature Review. J Cardiothorac Vasc Anesth. 2019 Sep;33(9):2525-2536. doi: 10.1053/j.jvca.2019.01.003. Epub 2019 Jan 4. PMID 30686657
- [Background] Kameda T, Mizuma Y, Taniguchi H, Fujita M, Taniguchi N. Point-of-care lung ultrasound for the assessment of pneumonia: a narrative review in the COVID-19 era. J Med Ultrason (2001). 2021 Jan;48(1):31-43. doi: 10.1007/s10396-020-01074-y. Epub 2021 Jan 13. PMID 33438132
- [Background] Mojoli F, Bouhemad B, Mongodi S, Lichtenstein D. Lung Ultrasound for Critically Ill Patients. Am J Respir Crit Care Med. 2019 Mar 15;199(6):701-714. doi: 10.1164/rccm.201802-0236CI. PMID 30372119
- [Background] Islam M, Levitus M, Eisen L, Shiloh AL, Fein D. Lung Ultrasound for the Diagnosis and Management of Acute Respiratory Failure. Lung. 2020 Feb;198(1):1-11. doi: 10.1007/s00408-019-00309-1. Epub 2020 Jan 1. PMID 31894411
- [Background] Staub LJ, Mazzali Biscaro RR, Kaszubowski E, Maurici R. Lung Ultrasound for the Emergency Diagnosis of Pneumonia, Acute Heart Failure, and Exacerbations of Chronic Obstructive Pulmonary Disease/Asthma in Adults: A Systematic Review and Meta-analysis. J Emerg Med. 2019 Jan;56(1):53-69. doi: 10.1016/j.jemermed.2018.09.009. Epub 2018 Oct 9. PMID 30314929
- [Background] Diaz-Gomez JL, Mayo PH, Koenig SJ. Point-of-Care Ultrasonography. N Engl J Med. 2021 Oct 21;385(17):1593-1602. doi: 10.1056/NEJMra1916062. No abstract available. PMID 34670045
- [Derived] Okoye C, Ticinesi A, Finazzi A, Bruni AA, Guarino D, Cerundolo N, Nouvenne A, Siniscalchi C, Meschi T, Lauretani F, Maggio M, Zucchini I, Torrini M, Cerasuolo M, Rizzo MR, Monzani F, Antonelli Incalzi R, Ungar A, Bellelli G, Scarlata S; GRETA research group on thoracic ultrasound in the older patient, Italian Society of Geriatrics and Gerontology (SIGG). Exploring the correlations of lung ultrasound with delirium and other clinical outcomes in older patients with respiratory failure admitted in acute geriatric units (ECO-AGE): protocol for a multicentre, prospective, observational study from the GRETA Group (Gruppo di Ricerca in Ecografia Toracica nell'Anziano) of the Italian Society of Gerontology and Geriatrics (SIGG). BMJ Open. 2025 Jul 28;15(7):e097229. doi: 10.1136/bmjopen-2024-097229. PMID 40721254